CLINICAL TRIAL: NCT00979654
Title: A Phase 2 Open-label Study to Evaluate the Long-term Safety of Sifalimumab in Adult Subjects With Systemic Lupus Erythematosus or Myositis
Brief Title: A Study to Evaluate the Long-Term Safety of MEDI-545 in Adult Participants With Systemic Lupus Erythematosus or Myositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP212
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Sifalimumab; MEDI-545
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — sifalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sifalimumab (MEDI-545) 500 or 600 milligram (mg) (Experimental): All participants will receive intravenous (IV) sifalimumab as fixed dose of 500 mg every 2 weeks (Q2W) on Day 1, Week 2, and Week 4, then every 4 weeks (Q4W) thereafter for a total of 156 weeks. The initial fixed dose of 500 mg is increased to 600 mg with subsequent protocol amendment.
  Interventions: Drug: Sifalimumab

INTERVENTIONS:
Drug: Sifalimumab — All participants will receive intravenous (IV) sifalimumab as fixed dose of 500 mg every 2 weeks (Q2W) on Day 1, Week 2, and Week 4, then every 4 weeks (Q4W) thereafter for a total of 156 weeks. The initial fixed dose of 500 mg is increased to 600 mg with subsequent protocol amendment.

SUMMARY:
The objective of this study is to assess the safety and tolerability of sifalimumab in adult participants with active systemic lupus erythematosus (SLE) or active dermatomyositis (DM) or polymyositis (PM) who participated in the following clinical studies: MI-CP151, MI-CP152, or MI-CP179.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the long-term safety and tolerability of multiple intravenous (IV) doses of sifalimumab in adult participants with active SLE or DM or PM who were previously treated with investigational product (sifalimumab or placebo) in one of the following sifalimumab clinical studies: MI-CP151, MI-CP152, or MI-CP179.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of screening.
* Written informed consent and any locally required authorization [example, Health Insurance Portability and Accountability Act (HIPAA) in the United States of America (USA), European Union (EU) Data Privacy Directive in the EU] obtained from the participant/legal representative prior to performing any protocol-related procedures, including Screening evaluations.
* Female participants of childbearing potential who are sexually active must use must use 2 effective methods of avoiding pregnancy from Screening, and must agree to continue using such precautions for 26 weeks after the final dose of investigational product.
* Males, unless surgically sterile, must use 2 effective methods of birth control with a female partner and must agree to continue using such contraceptive precautions from Screening until 26 weeks after the final dose of investigational product. If female, unless cervix has been surgically removed, have had a Pap smear with no evidence of malignancy within 6 months of baseline (defined as Day 1).
* Must have qualified for and received investigational product (sifalimumab or placebo) and completed the treatment period plus follow-up (through Day 266 for participants from MI-CP151 and MI-CP152 or through Day 168 for participants from MI-CP179) in one of the following sifalimumab clinical studies: MI-CP151, MI-CP152, or MI-CP179, ability to complete the study period through the final visit, willing to forego other forms of experimental drug treatment during the study.

Exclusion Criteria:

* Discontinued investigational product (sifalimumab) for safety reasons from any previous sifalimumab clinical study.
* For participants with systemic lupus erythematosus (SLE): Active severe or unstable neuropsychiatric SLE, that in the opinion of the investigator, would make the participant unsuitable for the study or unable to fully understand the informed consent, Active severe or unstable renal disease that in the opinion of the investigator would make the participant unsuitable for this study
* For participants with dermatomyositis (DM) or polymyositis (PM): Inclusion body myositis, cancer-associated myositis, myositis associated with another connective tissue disease, environmentally-associated myositis, or drug-related myopathy, a history of or a family history of non-inflammatory myopathy, scapular winging, atrophy, or hypertrophy of the calf muscles, Active Hepatitis A, confirmed positive tests for hepatitis B surface antigen (HbsAg) and hepatitis B core antibody (HbcAb) or hepatitis C serology. Isolated HbcAb positivity will be explored with additional reflex testing to determine eligibility.
* Evidence of active tuberculosis (TB), either treated or untreated, or latent TB without completion of an appropriate course of treatment or appropriate ongoing prophylactic treatment, history of severe viral infection, such as disseminated herpes, herpes encephalitis, or ophthalmic herpes.
* Any of the following medications within 6 months before entry into the study: Leflunomide greater than (>) 20 milligram/day, Cyclophosphamide (or any other alkylating agent).
* Any of the following medications within 28 days before entry into the study: Prednisone or equivalent > 30 mg/day or > 0.5 mg/kg, whichever is the lesser amount, Cyclosporine at any dose, Thalidomide at any dose, Interferon alpha 2b, Hydroxychloroquine > 600 mg/day, Mycophenolate mofetil > 3 gram/day, Methotrexate > 25 mg/week, Azathioprine > 3 mg/kilogram (kg)/day, Combination of leflunomide and methotrexate
* Nonstable doses of one or more of the following medications within 28 days before entry into the study: Hydroxychloroquine, Mycophenolate mofetil, Methotrexate, Azathioprine
* At Screening blood tests (within 28 days before entry into the study), any of the following: Total bilirubin > upper limit of normal (ULN), Neutrophil count < 1,500/microliter (mcl) (or < 1.5 × 109/L), Platelet count < 60,000/microliter (mcl) (or < 60 × 109/L), Hemoglobin (Hgb) < 7 gram per decilitre (g/dL) (or < 70 g/L).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Green, Study Director — MedImmune LLC
Locations (28):
- United States (24):
  - Research Site, Anniston, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, San Leandro, California
  - Research Site, Upland, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Ocala, Florida
  - Research Site, Tampa, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Cumberland, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Lake Success, New York
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Brazil (2):
  - Research Site, Curitiba
  - Research Site, São Paulo
- Research Site, Winnipeg, Manitoba, Canada
- Research Site, Santiago, Chile

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 118 participants were Screened out of which 15 participants did not meet eligibility criteria and were considered screen failures, and 103 participants were entered into the study.
Groups:
- MEDI-545: All participants received intravenous (IV) sifalimumab as fixed dose of 500 mg every 2 weeks (Q2W) on Day 1, Week 2, and Week 4, then every 4 weeks (Q4W) thereafter for a total of 156 weeks. The initial fixed dose of 500 mg was increased to 600 mg with subsequent protocol amendment.
Period: Overall Study
Arm/Group | MEDI-545
Started | 103
Completed | 67
Not Completed | 36
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 22
Not completed — Death | 1
Not completed — Lack of Efficacy | 6
Not completed — Adverse Event | 1
Not completed — Adverse Event of Diverticulitis | 1
Not completed — Per Principal Investigator's Discretion | 1
Not completed — Patient Wanted to Pursue Other Treatment | 1
Not completed — Serious Adverse Event | 1
Not completed — Unfavorable Risk-Benefit Analysis | 1

BASELINE CHARACTERISTICS:
Arm/Group | MEDI-545
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (9.9)
Age, Customized [Number; unit: Participants]
  < 40 | 21
  40 - <65 | 78
  >= 65 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received investigational product. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of investigational product and 30 days after the last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From start of study drug administration until week 182
Population: Safety Population included all participants who received at least one dose of investigational product.
Measure: Number; unit: participants
Groups:
- Sifalimumab (MEDI-545) 500 or 600 Milligram (mg): All participants received intravenous (IV) sifalimumab as fixed dose of 500 mg every 2 weeks (Q2W) on Day 1, Week 2, and Week 4, then every 4 weeks (Q4W) thereafter for a total of 156 weeks. The initial fixed dose of 500 mg was increased to 600 mg with subsequent protocol amendment.
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 103
participants
  TEAEs | 101
  TESAEs | 27

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Sifalimumab
Description: The Cmax is the maximum observed plasma concentration of sifalimumab.
Time Frame: Pre-infusion and End of Infusion on Day 1
Population: The PK Population included all participants who received at least one dose of investigational product and had at least one evaluable sifalimumab serum concentration. Here, "N" is number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 94
microgram per milliliter (mcg/mL) | 225.569 (78.842)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Sifalimumab
Description: The Tmax is the time to reach maximum observed plasma concentration of sifalimumab.
Time Frame: Pre-infusion and End of Infusion on Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 94
days | 0.049 [0.04 to 0.13]

4. Secondary Outcome: Time to Last Quantifiable Plasma Concentration (Tlast) of Sifalimumab
Description: The Tlast is the time to last quantifiable plasma concentration (Tlast) of sifalimumab.
Time Frame: Pre-infusion and End of Infusion on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 99
days | 14.413 (1.693)

5. Secondary Outcome: Minimum Observed Serum Concentration (Ctrough) of Sifalimumab
Description: The Ctrough is the minimum observed serum concentration of sifalimumab.
Time Frame: Pre-infusion and End of Infusion on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 99
mcg/mL | 65.009 (30.516)

6. Secondary Outcome: Area Under the Serum Concentration-time Curve Over the Dosing Interval (AUCtau) of Sifalimumab
Description: The AUCtau is the area under the serum concentration-time curve over the dosing interval of sifalimumab.
Time Frame: Pre-infusion and End of Infusion on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram.day per milliliter(mcg*day/mL)
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 93
microgram.day per milliliter(mcg*day/mL) | 2084.180 (665.882)

7. Secondary Outcome: Minimum Observed Serum Concentration at Steady State (Ctrough,ss) of Sifalimumab
Description: The Ctrough is the minimum observed serum concentration at steady state of sifalimumab.
Time Frame: Pre-infusion and End of Infusion on Day 1 and Week 2, 4, 8, 12, 24, 52, 104, 156 and 168
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 87
mcg/mL | 78.731 (53.942)

8. Secondary Outcome: Accumulation Index for Minimum Observed Serum Concentration (Ctrough) of Sifalimumab
Description: The Ctrough is the minimum observed serum concentration of sifalimumab. Accumulation Index is calculated as Ctrough value at steady state divided by Ctrough value after first dose.
Time Frame: Pre-infusion and End of Infusion on Day 1 and Week 2, 4, 8, 12, 24, 52, 104, 156 and 168
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 84
ratio | 1.217 (0.808)

9. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody
Description: Participants tested for immunogenicity to Sifalimumab (MEDI-545) from Day 1 to the end of study.
Time Frame: Day 1 and Week 12, 24, 52, 104, 156 and 168
Population: Safety Population included all participants who received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Sifalimumab (MEDI-545) 500 or 600 Milligram (mg)
Number analyzed (Participants) | 103
Participants
  Day 1 | 5
  Week 12 | 0
  Week 24 | 0
  Week 52 | 1
  Week 104 | 4
  Week 156 | 1
  Week 168 | 4
  Any Day Post Baseline | 9

ADVERSE EVENTS:
Time Frame: From start of study drug administration until week 182
Description: The safety Population included all participants who received at least one dose of investigational product.
Arm/Group | MEDI-545
Serious Adverse Events (participants affected / at risk) | 27/103
Other Adverse Events (participants affected / at risk) | 89/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-545 (N=103)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Bone abscess (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3)
Diverticulitis (Infections and infestations) | 2 (2)
Enteritis infectious (Infections and infestations) | 1 (1)
Herpes simplex meningitis (Infections and infestations) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-545 (N=103)
Abdominal pain (Gastrointestinal disorders) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 16 (24)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 20 (28)
Vomiting (Gastrointestinal disorders) | 11 (17)
Fatigue (General disorders) | 8 (9)
Seasonal allergy (Immune system disorders) | 7 (7)
Bronchitis (Infections and infestations) | 23 (36)
Gastroenteritis (Infections and infestations) | 7 (7)
Gastroenteritis viral (Infections and infestations) | 6 (10)
Herpes zoster (Infections and infestations) | 8 (8)
Influenza (Infections and infestations) | 7 (10)
Nasopharyngitis (Infections and infestations) | 22 (36)
Sinusitis (Infections and infestations) | 18 (38)
Upper respiratory tract infection (Infections and infestations) | 40 (65)
Urinary tract infection (Infections and infestations) | 30 (62)
Vulvovaginal mycotic infection (Infections and infestations) | 6 (13)
Contusion (Injury, poisoning and procedural complications) | 9 (12)
Fall (Injury, poisoning and procedural complications) | 6 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 7 (9)
Dizziness (Nervous system disorders) | 10 (14)
Headache (Nervous system disorders) | 22 (27)
Anxiety (Psychiatric disorders) | 7 (7)
Depression (Psychiatric disorders) | 9 (11)
Insomnia (Psychiatric disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 8 (12)
Hypertension (Vascular disorders) | 9 (12)

LIMITATIONS AND CAVEATS:
A business decision was made to discontinue the development of sifalimumab in favor of another type 1 interferon (IFN) inhibitor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.